CLINICAL TRIAL: NCT01590329
Title: A Proof of Concept Cases Series on the Use of the Epidermal Expansion System to Harvest and Place Suction Blister Epidermal Grafts on Hypopigmented Skin and Surgical Wounds
Brief Title: Use of Epidermal Expansion System for Epidermal Grafting on Hypopigmented Skin and Surgical Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Momelan Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMT-LSS-1
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Surgical Wound; Hypo-pigmented Skin
Keywords: Skin surgery; Micrografting; Hypo-pigmentation
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micrografting (Experimental)
  Interventions: Device: Momelan Technologies Epidermal Graft Harvesting System

INTERVENTIONS:
Device: Momelan Technologies Epidermal Graft Harvesting System — The procurement of the epidermal micro graft involves the use of MoMelan Technologies suction blister system, which consists of a control harvester. The device is applied to the subject's thigh to create blisters. The epidermal micrografts are then harvested and transferred to a commercially available sterile film dressing, placed on the surgical wound or prepared recipient site and the wound is then bandaged.

SUMMARY:
This case series will assess the use of suction blister epidermal grafts harvested by a novel device on select patients with hypo pigmented skin or surgical skin wounds.

DETAILED DESCRIPTION:
This study evaluates a novel micrografting technique to determine how it will influence the repigmentation of selected areas of hypopigmentation, and how it will influence the healing and pigmentation of surgical skin wounds. The Epidermal Expansion System (designed by MoMelan Technologies) will generate an array of small microblisters and transfer the micrografts to a sterile FDA cleared wound dressing for application to the subject's acute wound or prepared recipient site. The sponsor hypothesizes that applying expanded micrografts to target sites will result in rapid healing of acute wounds and in repigmentation of hypopigmented skin as well as and provide improved cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult subject between 18 and 99 years of age
* Subject having an area of hypopigmentation or surgical wound considered appropriate by physician to receive epidermal micro grafting
* Willingness to participate in study by evidence of informed consent

Exclusion Criteria:

* Female subjects self-reported to be breastfeeding, pregnant or planning to become pregnant during the course of the study.
* Subject showing clinical signs of infection
* Subjects currently on immunosuppressive medications, chemotherapy or cytotoxic agents
* Subject participation in another interventional study with potential exposure to an investigational drug or device within the past 30 days or planned entry into another investigational study within 90 days after entrance into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Wound healing/pigmentation | up to 12 weeks

SECONDARY OUTCOMES:
Patient Satisfaction | 6-12 weeks
Physician Satisfaction | 6-12 weeks
Incidence of adverse events | 6-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roy Geronemus, MD, Principal Investigator — Laser and Skin Surgery Center of New York
Locations (1):
- Laser and Skin Surgery Center of New York, New York, New York, United States